CLINICAL TRIAL: NCT03257358
Title: A 12-Month, Prospective, Multicenter, Two-cohort, Nonrandomized, Open-label Study in Adult Patients With Relapsing Multiple Sclerosis (RMS), to Investigate Changes in Immune Phenotype Biomarkers After Treatment With 0.5mg Fingolimod [FLUENT]
Brief Title: A Study of Immune Phenotype Biomarkers in Patients With Relapsing Multiple Sclerosis (RMS) After Treatment With 0.5mg Fingolimod
Acronym: FLUENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CFTY720DUS40
Record Dates: First submitted 2017-08-18; First posted 2017-08-22 (Actual); Results first posted 2020-07-21 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; RMS; Relapsing Multiple Sclerosis (RMS); Multiple Sclerosis; MS; Multiple Sclerosis (MS); Fingolimod; FLUENT; Immune Phenotype; adult; FTY720
MeSH Terms: conditions — Multiple Sclerosis | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Intervention Model Description: Two-cohort, non-randomized, open-label multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Other): RMS patients who were newly prescribed commercially available fingolimod 0.5mg per day
  Interventions: Drug: Fingolimod
- Cohort 2 (Other): RMS patients who had been on commercially available fingolimod 0.5mg per day continuously for ≥ 2 years
  Interventions: Drug: Fingolimod

INTERVENTIONS:
Drug: Fingolimod — Commercially available 0.5mg hard capsules, taken orally once per day

SUMMARY:
A study of immune phenotype biomarkers in patients with Relapsing Multiple Sclerosis (RMS) after treatment with 0.5mg fingolimod

DETAILED DESCRIPTION:
This study used a 2-cohort, nonrandomized, open-label, multicenter design. Cohort 1: The first cohort was to be comprised of approximately 200 patients with RMS, who were newly prescribed commercially available fingolimod 0.5 mg/day. Cohort 2: The second cohort was to be comprised of approximately 200 RMS patients who had been on commercially available fingolimod 0.5 mg/day continuously without interruption of treatment for at least ≥ 2 years. Patients from both cohorts were recruited simultaneously from up to 125 MS centers in the United States. Both cohorts ran concurrently. The study consisted of 2 periods: Screening (up to 4 weeks) and Treatment period from Baseline (end of screening period considered as Day 1) up to 12 months with visits conducted at 3,6 and 12 months with a 14 day follow-up post treatment..

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing forms of Multiple Sclerosis
* Patients who started commercially prescribed fingolimod therapy 0.5mg per day OR patients already on commercially prescribed fingolimod 0.5mg per day continuously for ≥ 2 years

Exclusion Criteria (per USPI):

* Patients who in the last 6 months experienced myocardial infarction, unstable angina, stroke, transient ischemic stroke, decompensated heart failure requiring hospitalization or Class III/IV heart failure
* History or presence of Mobitz Type II second-degree or third-degree atrioventricular block or sick sinus syndrome, unless patient had a functioning pacemaker
* Baseline QTc interval ≥ 500 msec
* Treatment with Class Ia or Class III anti-arrhythmic drugs
* Patients who had a hypersensitivity reaction to fingolimod or any of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Louisville, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Ocala, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Sunrise, Florida
  - Novartis Investigative Site, Vero Beach, Florida
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Suwanee, Georgia
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Lutherville, Maryland
  - Novartis Investigative Site, Foxborough, Massachusetts
  - Novartis Investigative Site, Lexington, Massachusetts
  - Novartis Investigative Site, Wellesley, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Owosso, Michigan
  - Novartis Investigative Site, Golden Valley, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Fair Lawn, New Jersey
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, Plainview, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Mooresville, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Westerville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, Port Royal, South Carolina
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Falls Church, Virginia
  - Novartis Investigative Site, Vienna, Virginia
  - Novartis Investigative Site, Kirkland, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Huntington, West Virginia
  - Novartis Investigative Site, Green Bay, Wisconsin
  - Novartis Investigative Site, Milwaukee, Wisconsin
  - Novartis Investigative Site, Neenah, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=558

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 165 patients were enrolled but only 163 were treated and included in the Safety Set
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 165 | 217
Never Received Treatment | 2 | 0
Completed | 94 | 183
Not Completed | 71 | 34
Not completed — Adverse Event | 25 | 12
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 12 | 4
Not completed — Non-compliance with fingolimod treatment | 4 | 2
Not completed — Physician Decision | 2 | 2
Not completed — Protocol Violation | 5 | 3
Not completed — Technical problems | 4 | 1
Not completed — Withdrawal by Subject | 8 | 3
Not completed — Withdrawal of informed consent | 9 | 5
Not completed — New therapy for study indication | 1 | 0
Not completed — No longer requires treatment | 0 | 1

BASELINE CHARACTERISTICS:
Population: There were 165 participants enrolled in the trial but 2 participants in Cohort 1 never received treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 163 | 217 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (10.72) | 48.9 (9.94) | 45.9 (10.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 158 | 285
  Male | 36 | 59 | 95
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 136 | 186 | 322
  Black | 22 | 22 | 44
  Asian | 0 | 3 | 3
  Native American | 1 | 2 | 3
  Unknown | 3 | 1 | 4
  Other | 1 | 3 | 4
Time from Multiple Sclerosis Diagnosis until study treamtent [Mean (Standard Deviation); unit: years] | 6.78 (7.984) | 12.94 (7.007) | 10.30 (8.033)
Number of Patients with Relaspses within the last year [Number; unit: Number of patients with relapse] — Population: Missing data for some participants
  Number of patients with relapse
    Number of patients with at least 1 relapse: number analyzed (Participants) | 162 | 215 | 377
    Number of patients with at least 1 relapse | 101 | 32 | 133
    Number of patients with no relapse: number analyzed (Participants) | 162 | 215 | 377
    Number of patients with no relapse | 61 | 183 | 244

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 6 in CD4+ Naive T Cells (CCR7+ CD45RA+)
Description: Blood samples (approximately 60-80 ml) were collected at specifiied visits for biomarker and hematology assessments. In Cohort 1 patients it was critical that the blood sample was collected prior to administration of fingolimod, first dose observation (FDO). A central laboratory was used for analysis of all specimens collected.
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 404.4 (273.56) | 3.4 (20.69)
  Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Month 6 n=97,156 | 7.6 (38.04) | 4.8 (23.52)
  Change from BL to Month 6, n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6, n=97,156 | -411.4 (273.31) | 0.8 (25.12)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -413.4, 95% CI 2-sided [-422.7 to -404.], Standard Error of Mean 4.7
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -0.2, 95% CI 2-sided [-3.9 to 3.6], Standard Error of Mean 1.91

2. Primary Outcome: Change From Baseline to Month 6 in CD4+ Central Memory T Cells (CCR7+CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 374.6 (216.36) | 16.3 (45.11)
  Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Month 6 n=97,156 | 19.6 (58.77) | 18.3 (42.89)
  Change from BL to Month 6, n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6, n=97,156 | -368.9 (218.40) | 1.1 (51.29)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -368.7, 95% CI 2-sided [-382.8 to 354.7], Standard Error of Mean 7.08
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -0.1, 95% CI 2-sided [-7.1 to 6.9], Standard Error of Mean 3.54

3. Primary Outcome: Change From Baseline to Month 6 in CD4+ Effector Memory T Cells (CCR7-CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 74.3 (43.56) | 22.8 (41.21)
  Month 6, n=97,156: number analyzed (Participants) | 97 | 156
  Month 6, n=97,156 | 18.2 (23.00) | 21.7 (33.28)
  Change from BL to Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6 n=97,156 | -51.5 (36.24) | -2.0 (31.86)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -52.1, 95% CI 2-sided [-57.2 to -46.9], Standard Error of Mean 2.58
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -3.1, 95% CI 2-sided [-7.6 to 1.4], Standard Error of Mean 2.27

4. Primary Outcome: Change From Baseline to Month 6 in CD4+ Th1 Cells (CXCR3+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,211: number analyzed (Participants) | 148 | 211
  Baseline (BL) n=148,211 | 53.8 (38.29) | 11.1 (31.90)
  Month 6 n=104,180: number analyzed (Participants) | 104 | 180
  Month 6 n=104,180 | 7.6 (15.12) | 11.7 (33.33)
  Change from BL to Month 6 n=104,180: number analyzed (Participants) | 104 | 180
  Change from BL to Month 6 n=104,180 | -43.6 (32.51) | -0.7 (14.38)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -43.6, 95% CI 2-sided [-46.9 to -40.3], Standard Error of Mean 1.67
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -0.7, 95% CI 2-sided [-3.0 to 1.7], Standard Error of Mean 1.18

5. Primary Outcome: Change From Baseline to Month 6 in CD4+ Th2 Cells (CCR4+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,212: number analyzed (Participants) | 148 | 212
  Baseline (BL) n=148,212 | 35.9 (30.06) | 1.1 (4.01)
  Month 6 n=104,181: number analyzed (Participants) | 104 | 181
  Month 6 n=104,181 | 1.7 (4.17) | 1.6 (5.55)
  Change from BL to Month 6 n=104,181: number analyzed (Participants) | 104 | 181
  Change from BL to Month 6 n=104,181 | -36.1 (32.42) | 0.5 (5.28)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -36.3, 95% CI 2-sided [-37.2 to -35.3], Standard Error of Mean 0.48
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.4, 95% CI 2-sided [-0.4 to 1.2], Standard Error of Mean 0.42

6. Primary Outcome: Change From Baseline to Month 6 in CD4+ Th17 Cells (CCR6+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,212: number analyzed (Participants) | 148 | 212
  Baseline (BL) n=148,212 | 55.5 (36.60) | 2.4 (5.96)
  Month 6 n=104,181: number analyzed (Participants) | 104 | 181
  Month 6 n=104,181 | 3.1 (8.38) | 2.8 (6.91)
  Change from BL to Month 6 n=104,181: number analyzed (Participants) | 104 | 181
  Change from BL to Month 6 n=104,181 | -53.2 (39.01) | 0.5 (6.77)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -53.2, 95% CI 2-sided [-55.1 to -51.3], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.4, 95% CI 2-sided [-0.7 to 1.4], Standard Error of Mean 0.51

7. Primary Outcome: Change From Baseline to Month 6 in CD8+ Naive T Cells (CCR7+CD45RA+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 150.9 (119.48) | 1.8 (8.87)
  Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Month 6 n=97,156 | 4.2 (22.00) | 3.3 (15.84)
  Change from BL to Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6 n=97,156 | -139.3 (113.25) | 1.2 (14.89)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -140.4, 95% CI 2-sided [-145.8 to -135.0], Standard Error of Mean 2.71
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.7, 95% CI 2-sided [-1.9 to 3.3], Standard Error of Mean 1.30

8. Primary Outcome: Change From Baseline to Month 6 in CD8+ Central Memory T Cells (CCR7+CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 93.1 (75.22) | 5.6 (14.85)
  Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Month 6 n=97,156 | 5.9 (16.42) | 6.1 (12.97)
  Change from BL to Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6 n=97,156 | -85.2 (67.95) | 0.0 (15.92)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -85.2, 95% CI 2-sided [-89.0 to -81.4], Standard Error of Mean 1.92
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.2, 95% CI 2-sided [-2.3 to 1.9], Standard Error of Mean 1.06

9. Primary Outcome: Change From Baseline to Month 6 in CD8+ Effector Memory T Cells (CCR7-CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 108.2 (93.28) | 63.8 (115.28)
  Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Month 6 n=97,156 | 55.4 (102.88) | 52.6 (40.76)
  Change from BL to Month 6 n=97,156: number analyzed (Participants) | 97 | 156
  Change from BL to Month 6 n=97,156 | -40.6 (103.03) | -12.5 (116.16)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -27.9, 95% CI 2-sided [-51.1 to -4.8], Standard Error of Mean 11.65
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -9.4, 95% CI 2-sided [-16.3 to -2.6], Standard Error of Mean 3.47

10. Primary Outcome: Change From Baseline to Month 6 in Naive B Lymphocytes (CD19+CD27-)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 201.1 (134.16) | 18.1 (33.79)
  Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Month 6 n=101,176 | 15.0 (10.50) | 17.8 (19.99)
  Change from BL to Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Change from BL to Month 6 n=101,176 | -181.4 (125.71) | -0.2 (36.61)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -181.2, 95% CI 2-sided [-183.3 to -179.0], Standard Error of Mean 1.07
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -0.8, 95% CI 2-sided [-4.1 to 2.5], Standard Error of Mean 1.66

11. Primary Outcome: Change From Baseline to Month 6 in Memory B Lymphocytes (CD19+CD27+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 61.8 (74.29) | 3.3 (22.58)
  Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Month 6 n=101,176 | 3.8 (6.24) | 4.0 (21.18)
  Change from BL to Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Change from BL to Month 6 n=101,176 | -55.1 (74.36) | 0.3 (6.40)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -55.2, 95% CI 2-sided [-56.5 to -53.9], Standard Error of Mean 0.66
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.3, 95% CI 2-sided [-0.5 to 1.1], Standard Error of Mean 0.42

12. Primary Outcome: Change From Baseline to Month 6 in Regulatory B Lymphocytes (CD19+CD24+CD38+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 12.3 (12.88) | 5.3 (7.66)
  Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Month 6 n=101,176 | 4.8 (3.92) | 6.1 (5.16)
  Change from BL to Month 6 n=101,176: number analyzed (Participants) | 101 | 176
  Change from BL to Month 6 n=101,176 | -7.4 (10.64) | 0.9 (8.15)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -7.2, 95% CI 2-sided [-8.0 to -6.4], Standard Error of Mean 0.40
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 1.1, 95% CI 2-sided [0.3 to 2.0], Standard Error of Mean 0.43

13. Primary Outcome: Change From Baseline to Month 6 in Monocytes (CD14+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=150,197: number analyzed (Participants) | 150 | 197
  Baseline (BL) n=150,197 | 329.6 (167.52) | 251.7 (118.46)
  Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Month 6 n=105,166 | 384.7 (148.76) | 379.2 (131.42)
  Change from BL to Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Change from BL to Month 6 n=105,166 | 66.1 (139.24) | 123.1 (123.85)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = 69.4, 95% CI 2-sided [42.1 to 96.7], Standard Error of Mean 13.78
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 117.0, 95% CI 2-sided [97.1 to 136.9], Standard Error of Mean 10.07

14. Primary Outcome: Change From Baseline to Month 6 in Neutrophils (CD16+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=149,197: number analyzed (Participants) | 149 | 197
  Baseline (BL) n=149,197 | 4041.4 (1576.73) | 3717.9 (1552.87)
  Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Month 6 n=105,166 | 3505.4 (1512.81) | 3312.6 (1311.04)
  Change from BL to Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Change from BL to Month 6 n=105,166 | -586.0 (1463.26) | -439.6 (1274.80)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -782.6, 95% CI 2-sided [-1058.2 to -507.1], Standard Error of Mean 138.90
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -485.9, 95% CI 2-sided [-667.3 to -304.4], Standard Error of Mean 91.88

15. Primary Outcome: Change From Baseline to Month 6 in NK Cells (CD56+)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=149,197: number analyzed (Participants) | 149 | 197
  Baseline (BL) n=149,197 | 166.4 (98.23) | 181.0 (113.95)
  Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Month 6 n=105,166 | 133.6 (83.41) | 154.5 (88.99)
  Change from BL to Month 6 n=105,166: number analyzed (Participants) | 105 | 166
  Change from BL to Month 6 n=105,166 | -29.4 (76.42) | -28.0 (81.73)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -33.3, 95% CI 2-sided [-48.2 to -18.5], Standard Error of Mean 7.47
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -25.8, 95% CI 2-sided [-36.7 to -14.9], Standard Error of Mean 5.52

16. Primary Outcome: Change From Baseline to Month 6 in Total CD4+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=156,213: number analyzed (Participants) | 156 | 213
  Baseline (BL) n=156,213 | 936.3 (443.31) | 64.4 (122.56)
  Month 6 n=110,182: number analyzed (Participants) | 110 | 182
  Month 6 n=110,182 | 53.4 (114.61) | 71.3 (112.50)
  Change from BL to Month 6 n=110,182: number analyzed (Participants) | 110 | 182
  Change from BL to Month 6 n=110,182 | -884.1 (440.65) | 1.4 (105.17)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -888.7, 95% CI 2-sided [-914.6 to -862.7], Standard Error of Mean 13.10
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -3.3, 95% CI 2-sided [-17.6 to 11.0], Standard Error of Mean 7.24

17. Primary Outcome: Change From Baseline to Month 6 in Total CD4+ Differential Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=157,213: number analyzed (Participants) | 157 | 213
  Baseline (BL) n=157,213 | 49.40 (10.115) | 11.95 (12.637)
  Month 6 n=111,183: number analyzed (Participants) | 111 | 183
  Month 6 n=111,183 | 11.08 (9.875) | 12.82 (13.687)
  Change from BL to Month 6 n=111,183: number analyzed (Participants) | 111 | 183
  Change from BL to Month 6 n=111,183 | -39.09 (12.052) | 0.32 (6.119)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -39.50, 95% CI 2-sided [-41.59 to -37.42], Standard Error of Mean 1.053
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.14, 95% CI 2-sided [-0.87 to 1.14], Standard Error of Mean 0.510

18. Primary Outcome: Change From Baseline to Month 6 in Total CD8+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=156,213: number analyzed (Participants) | 156 | 213
  Baseline (BL) n=156,213 | 419.9 (257.71) | 124.6 (213.41)
  Month 6 n=110,182: number analyzed (Participants) | 110 | 182
  Month 6 n=110,182 | 120.1 (148.82) | 116.8 (101.44)
  Change from BL to Month 6 n=110,182: number analyzed (Participants) | 110 | 182
  Change from BL to Month 6 n=110,182 | -266.2 (209.45) | -13.5 (205.59)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -248.9, 95% CI 2-sided [-278.7 to -219.2], Standard Error of Mean 15.00
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -9.9, 95% CI 2-sided [-25.1 to 5.4], Standard Error of Mean 7.71

19. Primary Outcome: Change From Baseline to Month 6 in Total CD8+ Differential Cell Counts (%)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=157,213: number analyzed (Participants) | 157 | 213
  Baseline (BL) n=157,213 | 21.86 (7.852) | 25.25 (14.406)
  Month 6 n=111,183: number analyzed (Participants) | 111 | 183
  Month 6 n=111,183 | 25.33 (14.998) | 24.99 (13.863)
  Change from BL to Month 6: number analyzed (Participants) | 111 | 183
  Change from BL to Month 6 | 4.63 (11.327) | -0.39 (4.528)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = 5.60, 95% CI 2-sided [3.13 to 8.08], Standard Error of Mean 1.249
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.04, 95% CI 2-sided [-0.68 to 0.76], Standard Error of Mean 0.364

20. Primary Outcome: Change From Baseline to Month 6 in Total CD19+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=151,213: number analyzed (Participants) | 151 | 213
  Baseline (BL) n=151,213 | 259.7 (167.94) | 21.4 (45.19)
  Month 6 n=106,179: number analyzed (Participants) | 106 | 179
  Month 6 n=106,179 | 19.5 (15.91) | 21.8 (34.75)
  Change from BL to Month 6 n=106,179: number analyzed (Participants) | 106 | 179
  Change from BL to Month 6 n=106,179 | -231.3 (153.49) | 0.1 (40.66)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -231.0, 95% CI 2-sided [-234.5 to -227.6], Standard Error of Mean 1.75
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = -0.3, 95% CI 2-sided [-5.2 to 4.5], Standard Error of Mean 2.45

21. Primary Outcome: Change From Baseline to Month 6 in Total CD19+ Differential Cell Count (%)
Description: as for outcome 1
Time Frame: Baseline to Month 6
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=152,213: number analyzed (Participants) | 152 | 213
  Baseline (BL) n=152,213 | 13.97 (7.245) | 4.81 (5.294)
  Month 6 n=107,180: number analyzed (Participants) | 107 | 180
  Month 6 n=107,180 | 5.38 (4.368) | 4.83 (5.236)
  Change from BL to Month 6 n=107,180: number analyzed (Participants) | 107 | 180
  Change from BL to Month 6 n=107,180 | -8.53 (6.723) | 0.23 (3.027)
Statistical Analysis 1: Comparison: Cohort 1; Test type: Other — Estimation; ANCOVA; least squares mean = -8.30, 95% CI 2-sided [-9.21 to -7.40], Standard Error of Mean 0.455
Statistical Analysis 2: Comparison: Cohort 2; Test type: Other — Estimation; ANCOVA; least squares mean = 0.32, 95% CI 2-sided [-0.17 to 0.82], Standard Error of Mean 0.251

22. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Naive T Cells (CCR7+CD45RA+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 404.4 (273.56) | 3.4 (20.69)
  Change from BL to Month 12 n=82,150: number analyzed (Participants) | 82 | 150
  Change from BL to Month 12 n=82,150 | -376.3 (277.23) | -0.8 (20.10)

23. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Central Memory T Cells (CCR7+CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 374.6 (216.36) | 16.3 (45.11)
  Change from BL to Month 12 n=83,150: number analyzed (Participants) | 83 | 150
  Change from BL to Month 12 n=83,150 | -356.8 (237.76) | 3.9 (55.06)

24. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Effector Memory T Cells (CCR7-CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 74.3 (43.56) | 22.8 (41.21)
  Change from BL to Month 12 n=83,150: number analyzed (Participants) | 83 | 150
  Change from BL to Month 12 n=83,150 | -50.4 (40.40) | -3.3 (30.24)

25. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Th1 Cells (CXCR3+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,211: number analyzed (Participants) | 148 | 211
  Baseline (BL) n=148,211 | 53.8 (38.29) | 11.1 (31.90)
  Change from BL to Month 12 n=88,175: number analyzed (Participants) | 88 | 175
  Change from BL to Month 12 n=88,175 | -42.3 (38.9) | -2.1 (15.04)

26. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Th2 Cells (CCR4+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,212: number analyzed (Participants) | 148 | 212
  Baseline (BL) n=148,212 | 35.9 (30.06) | 1.1 (4.01)
  Change from BL to Month 12: number analyzed (Participants) | 88 | 175
  Change from BL to Month 12 | -36.3 (34.63) | 0.4 (4.93)

27. Secondary Outcome: Change From Baseline to Month 12 in CD4+ Th17 Cells (CCR6+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=148,212: number analyzed (Participants) | 148 | 212
  Baseline (BL) n=148,212 | 55.5 (36.60) | 2.4 (5.96)
  Change from BL to Month 12 n=88,175: number analyzed (Participants) | 88 | 175
  Change from BL to Month 12 n=88,175 | -52.1 (41.20) | 0.5 (7.70)

28. Secondary Outcome: Change From Baseline to Month 12 in CD8+ Naive T Cells (CCR7+CD45RA+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 150.9 (119.48) | 1.8 (8.87)
  Change from BL to Month 12 n=83,150: number analyzed (Participants) | 83 | 150
  Change from BL to Month 12 n=83,150 | -126.3 (103.38) | 0.6 (10.24)

29. Secondary Outcome: Change From Baseline to Month 12 in CD8+ Central Memory T Cells (CCR7+CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 93.1 (75.22) | 5.6 (14.85)
  Change from BL to Month 12 n=83,150: number analyzed (Participants) | 83 | 150
  Change from BL to Month 12 n=83,150 | -86.5 (75.75) | 0.0 (16.88)

30. Secondary Outcome: Change From Baseline to Month 12 in CD8+ Effector Memory T Cells (CCR7-CD45RA-CD45RO+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=147,188: number analyzed (Participants) | 147 | 188
  Baseline (BL) n=147,188 | 108.2 (93.28) | 63.8 (115.28)
  Change from BL to Month 12 n=83,150: number analyzed (Participants) | 83 | 150
  Change from BL to Month 12 n=83,150 | -55.9 (57.48) | -15.9 (122.31)

31. Secondary Outcome: Change From Baseline to Month 12 in Naive B Lymphocytes (CD19+CD27-)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 201.11 (134.16) | 18.1 (33.79)
  Change from BL to Month 12 n=82,174: number analyzed (Participants) | 82 | 174
  Change from BL to Month 12 n=82,174 | -177.0 (114.43) | -0.5 (40.72)

32. Secondary Outcome: Change From Baseline to Month 12 in Memory B Lymphocytes (CD19+CD27+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 61.8 (74.29) | 3.3 (22.58)
  Change from BL to Month 12 n=82,174: number analyzed (Participants) | 82 | 174
  Change from BL to Month 12 n=82,174 | -46.4 (39.15) | 1.4 (19.59)

33. Secondary Outcome: Change From Baseline to Month 12 in Regulatory B Lymphocytes (CD19+CD24+CD38+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=144,212: number analyzed (Participants) | 144 | 212
  Baseline (BL) n=144,212 | 12.3 (12.88) | 5.3 (7.66)
  Change from BL to Month 12 n=82,174: number analyzed (Participants) | 82 | 174
  Change from BL to Month 12 n=82,174 | -7.7 (11.60) | 0.8 (8.88)

34. Secondary Outcome: Change From Baseline to Month 12 in Monocytes (CD14+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=150,197: number analyzed (Participants) | 150 | 197
  Baseline (BL) n=150,197 | 329.6 (167.52) | 251.7 (118.46)
  Change from BL to Month 12 n=86,164: number analyzed (Participants) | 86 | 164
  Change from BL to Month 12 n=86,164 | 57.1 (139.91) | 112.4 (130.82)

35. Secondary Outcome: Change From Baseline to Month 12 in Neutrophils (CD16+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=149,197: number analyzed (Participants) | 149 | 197
  Baseline (BL) n=149,197 | 4041.4 (1576.73) | 3717.9 (1552.87)
  Change from BL to Month 12 n=87, 164: number analyzed (Participants) | 87 | 164
  Change from BL to Month 12 n=87, 164 | -815.9 (1368.23) | -345.0 (1253.29)

36. Secondary Outcome: Change From Baseline to Month 12 in NK Cells (CD56+)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=149,197: number analyzed (Participants) | 149 | 197
  Baseline (BL) n=149,197 | 166.4 (98.23) | 181.0 (113.95)
  Change from BL to Month 12 n=87,164: number analyzed (Participants) | 87 | 164
  Change from BL to Month 12 n=87,164 | -32.6 (97.86) | -28.9 (86.71)

37. Secondary Outcome: Change From Baseline to Month 12 in Total CD4+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=156,213: number analyzed (Participants) | 156 | 213
  Baseline (BL) n=156,213 | 936.3 (443.31) | 64.4 (122.56)
  Change from BL to Month 12 n=94,176: number analyzed (Participants) | 94 | 176
  Change from BL to Month 12 n=94,176 | -844.9 (439.92) | 0.7 (101.82)

38. Secondary Outcome: Change From Baseline to Month 12 in Total CD4+ Differential Cell Count (%)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=157,213: number analyzed (Participants) | 157 | 213
  Baseline (BL) n=157,213 | 49.40 (10.115) | 11.95 (12.637)
  Change from BL to Month 12 n=95,176: number analyzed (Participants) | 95 | 176
  Change from BL to Month 12 n=95,176 | -37.90 (12.756) | 0.70 (6.127)

39. Secondary Outcome: Change From Baseline to Month 12 in Total CD8+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=156,213: number analyzed (Participants) | 156 | 213
  Baseline (BL) n=156,213 | 419.9 (257.71) | 124.6 (213.41)
  Change from BL to Month 12 n=94,176: number analyzed (Participants) | 94 | 176
  Change from BL to Month 12 n=94,176 | -265.1 (168.81) | -11.6 (216.00)

40. Secondary Outcome: Change From Baseline to Month 12 in Total CD8+ Differential Cell Counts (%)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=157,213: number analyzed (Participants) | 157 | 213
  Baseline (BL) n=157,213 | 21.86 (7.852) | 25.25 (14.406)
  Change from BL to Month 12 n=95,176: number analyzed (Participants) | 95 | 176
  Change from BL to Month 12 n=95,176 | 4.33 (11.185) | 0.34 (5.150)

41. Secondary Outcome: Change From Baseline to Month 12 in Total CD19+ Absolute Cell Count
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=151,213: number analyzed (Participants) | 151 | 213
  Baseline (BL) n=151,213 | 259.7 (167.94) | 21.4 (45.19)
  Change from BL to Month 12 n=88,176: number analyzed (Participants) | 88 | 176
  Change from BL to Month 12 n=88,176 | -218.9 (127.69) | 1.0 (52.35)

42. Secondary Outcome: Change From Baseline to Month 12 in Total CD19+ Differential Cell Count (%)
Description: as for outcome 1
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=152,213: number analyzed (Participants) | 152 | 213
  Baseline (BL) n=152,213 | 13.97 (7.245) | 4.81 (5.294)
  Change from BL to Month 12 n=89,176: number analyzed (Participants) | 89 | 176
  Change from BL to Month 12 n=89,176 | -8.86 (7.222) | 0.20 (3.210)

43. Secondary Outcome: Multiple Sclerosis (MS) Relapses During Treatment
Description: A relapse is defined as the appearance of a new neurological abnormality or worsening of previously stable or improving pre-existing neurological abnormality, separated by at least 30 days from onset of a preceding clinical demyelinating event. The abnormality must be present for at least 24 hours and occur in the absence of fever (<37.5°C) or infection.
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Number; unit: relapses
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
relapses
  Number of patients with relapses | 11 | 13
  Total number of relapses | 12 | 13
  Relapses not requiring steroid use | 5 | 5
  Relapses requiring steroid use | 7 | 8
  Mild relapse | 5 | 8
  Moderate relapse | 6 | 5
  Severe relapse | 1 | 0

44. Secondary Outcome: Number of Participants Who Received Steroid Treatment for MS Relapses During Treatment
Description: as for outcome 43
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
Participants
  Patients with ≥ 1 relapses | 11 | 13
  Patients with relapse who received ≥ 1 steroid | 7 | 8
  Corticosteroids for systemic use | 7 | 8
  Methylprednisolone sodium succinate | 4 | 4
  Methylprednisolone | 3 | 2
  Prednisone | 0 | 3

45. Secondary Outcome: Change From Baseline in Patient Determined Disease Steps (PDDS)
Description: PDDS scoring ranges 0 to 8. 0 = Normal; 1 = Mild disability; 2 = Moderate disability; 3 = Gait disability; 4 = Early cane; 5 = Late cane; 6 = Bilateral support; 7 = Wheelchair/scooter; 8 = Bedridden.
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: scores
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
scores
  Baseline (BL) n=163,217 | 1.7 (1.85) | 1.8 (1.90)
  Month 12 n=103,188: number analyzed (Participants) | 103 | 188
  Month 12 n=103,188 | 1.8 (1.95) | 1.8 (2.02)
  Change from BL to Month 12 n=103,188: number analyzed (Participants) | 103 | 188
  Change from BL to Month 12 n=103,188 | -0.1 (0.87) | -0.0 (0.78)

46. Secondary Outcome: Change From Baseline in T2 Lesion Burden
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
number of lesions
  Baseline (BL) n=91,84: number analyzed (Participants) | 91 | 84
  Baseline (BL) n=91,84 | 8.1 (12.74) | 9.7 (15.47)
  Month 12 n=21,17: number analyzed (Participants) | 21 | 17
  Month 12 n=21,17 | 6.5 (8.20) | 13.1 (13.22)
  Change from BL to Month 12 n=21,17: number analyzed (Participants) | 21 | 17
  Change from BL to Month 12 n=21,17 | -0.8 (2.36) | 3.2 (12.46)

47. Secondary Outcome: Change From Baseline for New Gd-Enhancing T1 Lesion Count
Time Frame: Baseline to Month 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: number of lesions
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
number of lesions
  Baseline (BL) n=125,147: number analyzed (Participants) | 125 | 147
  Baseline (BL) n=125,147 | 0.4 (1.09) | 0.2 (1.21)
  Month 12 n=33,28: number analyzed (Participants) | 33 | 28
  Month 12 n=33,28 | 0.1 (0.24) | 0.2 (0.83)
  Change from BL to Month 12 n=33,28: number analyzed (Participants) | 33 | 28
  Change from BL to Month 12 n=33,28 | -0.2 (0.61) | 0.2 (0.77)

48. Secondary Outcome: Change From Baseline to Months 6 and 12 in the Anti-JCV Antibody Index (Index/Value)
Time Frame: Baseline to Month 6 and 12
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 163 | 217
cells/uL
  Baseline (BL) n=159,215: number analyzed (Participants) | 159 | 215
  Baseline (BL) n=159,215 | 1.273 (1.2930) | 1.391 (1.2600)
  Change from BL to Month 6 n=116,195: number analyzed (Participants) | 116 | 195
  Change from BL to Month 6 n=116,195 | 0.038 (0.2874) | 0.045 (0.4724)
  Change from BL to Month 12 n=100,180: number analyzed (Participants) | 100 | 180
  Change from BL to Month 12 n=100,180 | 0.040 (0.3397) | 0.145 (0.6062)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 18. 5 months
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/163 | 0/217
Serious Adverse Events (participants affected / at risk) | 9/163 | 12/217
Other Adverse Events (participants affected / at risk) | 70/163 | 66/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=163) | Cohort 2 (N=217)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Hyperplasia (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Histoplasmosis disseminated (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Multiple sclerosis relapse (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=163) | Cohort 2 (N=217)
Leukopenia (Blood and lymphatic system disorders) | 3 | 2
Lymphopenia (Blood and lymphatic system disorders) | 9 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Bradycardia (Cardiac disorders) | 2 | 0
Blepharospasm (Eye disorders) | 2 | 0
Diplopia (Eye disorders) | 2 | 0
Eye pain (Eye disorders) | 2 | 0
Macular oedema (Eye disorders) | 2 | 0
Photopsia (Eye disorders) | 2 | 0
Vision blurred (Eye disorders) | 2 | 0
Visual impairment (Eye disorders) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Chest discomfort (General disorders) | 3 | 0
Fatigue (General disorders) | 8 | 3
Gait disturbance (General disorders) | 3 | 3
Acute sinusitis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 8 | 6
Urinary tract infection (Infections and infestations) | 0 | 7
Fall (Injury, poisoning and procedural complications) | 5 | 12
Alanine aminotransferase increased (Investigations) | 2 | 3
Aspartate aminotransferase increased (Investigations) | 2 | 3
Lymphocyte count decreased (Investigations) | 2 | 2
Transaminases increased (Investigations) | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 3
Carpal tunnel syndrome (Nervous system disorders) | 3 | 0
Central nervous system lesion (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 6 | 1
Headache (Nervous system disorders) | 13 | 4
Hypoaesthesia (Nervous system disorders) | 5 | 1
Migraine (Nervous system disorders) | 5 | 1
Paraesthesia (Nervous system disorders) | 3 | 2
Tremor (Nervous system disorders) | 4 | 0
Trigeminal neuralgia (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 5 | 3
Depression (Psychiatric disorders) | 5 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Hypertension (Vascular disorders) | 4 | 4
Hypotension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT03257358/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03257358/SAP_001.pdf